CLINICAL TRIAL: NCT04475133
Title: Effects of Percutaneous Neuromodulation on Plasticity in the Somatosensory System
Brief Title: Effects of Percutaneous Neuromodulation on Plasticity in the Somatosensory System in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Francisco Ortega Rehabilitacion Avanzada SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMP19/20-FREMPI
Record Dates: First submitted 2020-07-08; First posted 2020-07-17 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Echography guided percutaneous neuromodulation; Plasticity; somatomotor system; Peripheral nerve stimulation; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized intervention of repeated measures, quadruple-blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Order of treatments was randomized by a third person not involved in any of the other phases. Also, after the care provider has inserted the needle in the three groups, another third person without involvement in any other phase of the study choose the assigned treatment between three pre-programmed closed set of parameters in the stimulation machine, thus leaving treatment unknown for the care provider, the participant, the investigator and the outcome assessor, which received only encoded names for the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-frequency and high-intensity (Experimental): The intervention of ultrasound guided percutaneous neuromodulation is applied over the median nerve.
  The parameters are continuous stimulation of low frequency (2 hz) and high intensity (slightly painful) during 16 minutes.
  Interventions: Other: Ultrasound guided percutaneous neuromodulation
- High-frequency and low-intensity (Experimental): The intervention of ultrasound guided percutaneous neuromodulation is applied over the median nerve.
  The parameters are high frequency (100 hz) and low intensity trains. There are 5 trains, 5 second active current and 55 second without current per train.
  The current is off on the first 11 minutes and the next 5 minutes it will be on. The total time is 16 minutes.
  Interventions: Other: Ultrasound guided percutaneous neuromodulation
- Control group (Sham Comparator): The intervention of ultrasound guided percutaneous neuromodulation is applied over the median nerve without current during 16 minutes.
  Interventions: Other: Ultrasound guided percutaneous neuromodulation

INTERVENTIONS:
Other: Ultrasound guided percutaneous neuromodulation — It is a technique that consists in the electrical stimulation of peripheral nerve trunks, inserting an acupuncture needle in its path and using it as an electrode to apply electrical current

SUMMARY:
Echography guided percutaneous neuromodulation is a physical therapy technique, whose main objective is the treatment of pain with direct stimulation of the peripheral nerves using a rome needle of acupuncture as an active electrode for applying currents of electrostimulation.

The neurophysiological basis and the effects on the sensory and motor systems of this technique are not characterised. The present study proposes to perform the intervention on the area adjacent to the median nerve and to apply different stimulation protocols on healthy subjects to answer those questions.

DETAILED DESCRIPTION:
Intervention is going to be performed in the medial side of the arm, where the median nerve is accessible to the intervention. The theoretical basis of the technique is to produce specific controlled changes in the somatosensory system using synaptic plasticity, to ultimate affect the perception of pain through reduction of nociception afference. Subsequently, the protocols are based on synaptic physiology and the circuitry of the somatosensory system.

The protocols are the following:

1. - low-frequency and high-intensity of stimulation: 2hz during 16 min at an slightly annoying intensity, to induce synaptic depression on the c-fibers circuit, presumably carrying nociception.
2. - high-frequency and low-intensity of stimulation: 100 hz in 5 second trains, separated by 1 min of no current with a perceptible but mild intensity, to induce potentiation of a-beta fibers, presumably englobing mechanoreceptors which inhibit nociception through gate control in the spinal cord.
3. - placebo group has got the same intervention, but without current.

The study design is an experimental clinical trial, with randomized order of intervention with repeated measurements. This means each subject is having the three protocols at randomized order, with a gap of at least two weeks between them. The study is triple-blinded.

Somatomotor system variables, as sensory and pain pressure thresholds, grip strength, surface electromyographic activity and blood flow are evaluated on the hand of the subject. The arm to treat was also randomized for each subject The measurements are pre-intervention, post-intervention and 24 hours after the intervention for each protocol. Blood flow are measured only pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion criteria:

* healthy.
* more than 18 years old
* amateur athlete.

Exclusion criteria:

* to suffer or to have suffered any pathology on the arm on the last 30 days.
* to suffer some disease discouraging current application or needle¡ing, as coagulation deficit, etc.
* to suffer some disease as diabetes mellitus, cancer, neurology disease, depression, fibromyalgia, etc.
* to consume drugs as coagulants, anti-depressant, pregabalin, etc during investigation or the first week before investigation.
* to consume nsaids the last 48 hours before investigation or during investigation.
* to consume opioids the first week before investigation or during investigation.
* belonephobia.
* professional athlete
* to be pregnant
* to suffer immunodepression

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Mechanical Threshold elicited with Von Frey Filaments | Pre-intervention / baseline
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of mechanical sensation, that caliber is considered the pressure threshold to elicit mechanical. The test is performed with subject's eyes closed
Mechanical Threshold elicited with Von Frey Filaments | Immediately after the intervention
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of mechanical sensation, that caliber is considered the pressure threshold to elicit mechanical. The test is performed with subject's eyes closed.
Mechanical Threshold elicited with Von Frey Filaments | 24 hours after the intervention
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of mechanical sensation, that caliber is considered the pressure threshold to elicit mechanical. The test is performed with subject's eyes closed.
Pinprick pain threshold elicited with Von Frey Filaments | pre-intervention / baseline
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of pinprick sensation, that caliber is considered the pressure threshold to elicit pinprick pain. The test is performed with subject's eyes closed
Pinprick pain threshold elicited with Von Frey Filaments | Immediately after the intervention
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of pinprick sensation, that caliber is considered the pressure threshold to elicit pinprick pain. The test is performed with subject's eyes closed
Pinprick pain threshold elicited with Von Frey Filaments | 24 hours after the intervention
  We use Von Frey Filaments of increasing caliber to make pression in the evaluated areas. When the test subject reports perception of pinprick sensation, that caliber is considered the pressure threshold to elicit pinprick pain. The test is performed with subject's eyes closed
Pain evocated with Von Frey Filaments. | Pre-intervention / baseline
  We use Von Frey Filaments of increasing caliber to make pression with 100g, 180g and 300g in the evaluated areas. Each filament to make pression three times. The subject reports the pain in a scale of 0-10 number (scale NSR: 0 is any pain and 10 is the maximal perception of pain. The test is performed with subject's eyes closed.
Pain evocated with Von Frey Filaments. | Immediately after the intervention
  We use Von Frey Filaments of increasing caliber to make pression with 100g, 180g and 300g in the evaluated areas. Each filament to make pression three times. The subject reports the pain in a scale of 0-10 number (scale NSR: 0 is any pain and 10 is the maximal perception of pain. The test is performed with subject's eyes closed.
Pain evocated with Von Frey Filaments. | 24 hours after the intervention
  We use Von Frey Filaments of increasing caliber to make pression with 100g, 180g and 300g in the evaluated areas. Each filament to make pression three times. The subject reports the pain in a scale of 0-10 number (scale NSR: 0 is any pain and 10 is the maximal perception of pain. The test is performed with subject's eyes closed.
Pressure pain threshold with algometer. | pre-intervention / baseline
  On the marked areas we make pressure with pressure algometer. When the subject experiences any sense of pain, he/she has to say "stop" and immediately the algometer was removed. The number in Kg marked by the algometer is annotated. The mean of two measurements was taken for analysis. The second measurement was taken with a minimum of 30 seconds after the previous one.
Change in pressure pain threshold with algometer. | Immediately after the intervention
  On the marked areas we make pressure with pressure algometer. When the subject experiences any sense of pain, he/she has to say "stop" and immediately the algometer was removed. The number in Kg marked by the algometer is annotated. The mean of two measurements was taken for analysis. The second measurement was taken with a minimum of 30 seconds after the previous one.
Change in pressure pain threshold with algometer. | 24 hours after the intervention
  On the marked areas we make pressure with pressure algometer. When the subject experiences any sense of pain, he/she has to say "stop" and immediately the algometer was removed. The number in Kg marked by the algometer is annotated. The mean of two measurements was taken for analysis. The second measurement was taken with a minimum of 30 seconds after the previous one.
Maximum grip force with dynamometer | pre-intervention / baseline
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Change in maximum grip force with dynamometer | Immediately after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Change in maximum grip force with dynamometer. | 24 hours after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Maximum grip force with surface electromyography. | pre-intervention / baseline
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Change in maximum grip force with surface electromyography. | Immediately after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Change in maximum grip force with surface electromyography. | 24 hours after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during 5 second, 3 times with 30 seconds to rest between them.
Arterial peak systolic velocity with Color Doppler Ultrasonography | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial peak systolic during 5 cardiac cycles.
Change in arterial peak systolic velocity with Color Doppler Ultrasonography in placebo group | Immediately after the needle insertion
  In placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial peak systolic during 5 cardiac cycles inmediately after introduce the needly in the arm.
Change in arterial peak systolic velocity with Color Doppler Ultrasonography | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial peak systolic during 5 cardiac cycles.
Arterial volume flow with Color Doppler Ultrasonography | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial volume flow during 5 cardiac cycles.
Change in arterial volume flow with Color Doppler Ultrasonography | Immediately after the needle insertion
  In placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial volume flow during 5 cardiac cycles.
Change in arterial volume flow with Color Doppler Ultrasonography | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial volume flow during 5 cardiac cycles.

SECONDARY OUTCOMES:
Electric current threshold of perception with low frequency | pre-intervention / baseline
  Using the intervention needle as an active electrode. The parameters are 2 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Change in Electric current threshold of perception with low frequency | Immediately after the intervention
  Using the intervention needle as an active electrode. The parameters are 2 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Change in Electric current threshold of perception with low frequency | 24 hours after the intervention
  Using the intervention needle as an active electrode. The parameters are 2 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Electric current threshold of perception with high frequency | pre-intervention / baseline
  Using the intervention needle as an active electrode. The parameters are 100 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Change electric current threshold of perception with high frequency | Immediately after the intervention
  Using the intervention needle as an active electrode. The parameters are 100 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Change electric current threshold of perception with high frequency | 24 hours after the intervention
  Using the intervention needle as an active electrode. The parameters are 100 hz and 150 msec of pulse duration and the intensity was increased progressively. When the subject experienced any sense of pain, sensitivity and muscle contraction in the needle and arm, he/she must tell it and the threshold is annotated.
Force grip resistance with dynamometer | Pre-intervention / Baseline
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Change in Force grip resistance with dynamometer. | Immediately after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Change in Force grip resistance with dynamometer. | 24 hours after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Force grip resistance with surface electromyography. | Pre-intervention / Baseline
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Change in Force grip resistance with surface electromyography. | Immediately after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Change in Force grip resistance with surface electromyography. | 24 hours after the intervention
  The subject is standing with the dynamometer in his hand. He/she must press the dynamometer during one minute trying to maintain maximal force.
Neural tension test (ROM) | pre-intervention / baseline
  The subject is lying on the stretcher. We make a neurodynamic test and when she/he experience tension in his/her arm, she/he must tell us "stop". We measure the range of motion of the elbow extension as the outcome
Change in neural tension test (ROM) | Immediately after the intervention
  The subject is lying on the stretcher. We make a neurodynamic test and when she/he experience tension in his/her arm, she/he must tell us "stop". We measure the range of motion of the elbow extension as the outcome
Change in neural tension test (ROM) | 24 hours after the intervention
  The subject is lying on the stretcher. We make a neurodynamic test and when she/he experience tension in his/her arm, she/he must tell us "stop". We measure the range of motion of the elbow extension as the outcome
Change in arterial end-diastolic velocity with Color Doppler Ultrasonography | Immediately after the needle insertion
  In the placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial end-diastolic velocity during 5 cardiac cycles.
Arterial time average mean velocity during cardiac cycle with Color Doppler Ultrasonography | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average mean velocity during 5 cardiac cycles.
Change in arterial time average mean velocity during cardiac cycle with Color Doppler Ultrasonography | Immediately after the needle insertion
  In the placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average mean velocity during 5 cardiac cycles.
Arterial end-diastolic velocity with Color Doppler Ultrasonography | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial end-diastolic velocity during 5 cardiac cycles.
Change in arterial end-diastolic velocity with Color Doppler Ultrasonography | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial end-diastolic velocity during 5 cardiac cycles.
Change in arterial time average mean velocity during cardiac cycle with Color Doppler | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average mean velocity during 5 cardiac cycles.
Arterial time average maximun velocity during cardiac cycle with Color Doppler | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average maximun velocity during 5 cardiac cycles.
Change in arterial time average maximun velocity during cardiac cycle with Color Doppler | Immediately after the needle insertion
  In placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average maximun velocity during 5 cardiac cycles.
Change in arterial time average maximun velocity during cardiac cycle with Color Doppler | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial time average maximun velocity during 5 cardiac cycles.
Arterial pulsatility index during cardiac cycle with Color Doppler | pre-intervention / baseline
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial pulsatility index during 5 cardiac cycles.
Change in arterial pulsatility index during cardiac cycle with Color Doppler | Immediately after the needle insertion
  In placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial pulsatility index during 5 cardiac cycles.
Change in arterial pulsatility index during cardiac cycle with Color Doppler | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial pulsatility index during 5 cardiac cycles.
Arterial arterial resistivity index during cardiac cycle with Color Doppler | pre-intervention / baseline
  In placebo group, on the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial resistivity index during 5 cardiac cycles.
Change in arterial resistivity index during cardiac cycle with Color Doppler | Immediately after the needle insertion
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial resistivity index during 5 cardiac cycles.
Change in arterial resistivity index during cardiac cycle with Color Doppler | Immediately after the intervention
  On the marked areas (Brachial ipsilateral and contralateral, radial and ulnar arteries) we measure the arterial resistivity index during 5 cardiac cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Beltrá López, Principal Investigator — Clínica Francisco Javier Ortega Puebla
Locations (1):
- Clínica Francisco Ortega Rehabilitación Avanzada, S.L., Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson RD, Harris MA, Gunzler DD, Bennett ME, Chae J. Percutaneous peripheral nerve stimulation for chronic pain in subacromial impingement syndrome: a case series. Neuromodulation. 2014 Dec;17(8):771-6; discussion 776. doi: 10.1111/ner.12152. Epub 2014 Feb 11. PMID 24512114
- [Background] Toprak U, Selvi NA, Ates A, Erhuner Z, Bostanoglu S, Karademir MA, Karaaslan Y. Dynamic Doppler evaluation of the hand arteries of the patients with Raynaud's disease. Clin Rheumatol. 2009 Jun;28(6):679-83. doi: 10.1007/s10067-009-1131-1. Epub 2009 Feb 24. PMID 19238503
- [Result] Barlas P, Ting SL, Chesterton LS, Jones PW, Sim J. Effects of intensity of electroacupuncture upon experimental pain in healthy human volunteers: a randomized, double-blind, placebo-controlled study. Pain. 2006 May;122(1-2):81-9. doi: 10.1016/j.pain.2006.01.012. Epub 2006 Mar 9. PMID 16527396
- [Result] Bliss TV, Collingridge GL. A synaptic model of memory: long-term potentiation in the hippocampus. Nature. 1993 Jan 7;361(6407):31-9. doi: 10.1038/361031a0. PMID 8421494
- [Result] Bliss TV, Lomo T. Long-lasting potentiation of synaptic transmission in the dentate area of the anaesthetized rabbit following stimulation of the perforant path. J Physiol. 1973 Jul;232(2):331-56. doi: 10.1113/jphysiol.1973.sp010273. PMID 4727084
- [Result] Borg-Stein J, Simons DG. Focused review: myofascial pain. Arch Phys Med Rehabil. 2002 Mar;83(3 Suppl 1):S40-7, S48-9. doi: 10.1053/apmr.2002.32155. PMID 11973695
- [Result] Chae J, Wilson RD, Bennett ME, Lechman TE, Stager KW. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case series. Pain Pract. 2013 Jan;13(1):59-67. doi: 10.1111/j.1533-2500.2012.00541.x. Epub 2012 Mar 26. PMID 22448759
- [Result] Chapman CR, Gavrin J. Suffering: the contributions of persistent pain. Lancet. 1999 Jun 26;353(9171):2233-7. doi: 10.1016/S0140-6736(99)01308-2. PMID 10393002
- [Result] Chan AW, MacFarlane IA, Bowsher D, Campbell JA. Weighted needle pinprick sensory thresholds: a simple test of sensory function in diabetic peripheral neuropathy. J Neurol Neurosurg Psychiatry. 1992 Jan;55(1):56-9. doi: 10.1136/jnnp.55.1.56. PMID 1312581
- [Result] Corneil BD, Goonetilleke SC, Peel TR, Green KA, Welch ID. Ultrasound-guided insertion of intramuscular electrodes into suboccipital muscles in the non-human primate. J Electromyogr Kinesiol. 2012 Aug;22(4):553-9. doi: 10.1016/j.jelekin.2012.02.014. Epub 2012 Mar 22. PMID 22445030
- [Result] Dommerholt J. Dry needling - peripheral and central considerations. J Man Manip Ther. 2011 Nov;19(4):223-7. doi: 10.1179/106698111X13129729552065. PMID 23115475
- [Result] Domingo A, Mayoral O, Monterde S, Santafe MM. Neuromuscular damage and repair after dry needling in mice. Evid Based Complement Alternat Med. 2013;2013:260806. doi: 10.1155/2013/260806. Epub 2013 Apr 9. PMID 23662122
- [Result] Dubuisson D. Effect of dorsal-column stimulation on gelatinosa and marginal neurons of cat spinal cord. J Neurosurg. 1989 Feb;70(2):257-65. doi: 10.3171/jns.1989.70.2.0257. PMID 2913223
- [Result] Falowski S, Celii A, Sharan A. Spinal cord stimulation: an update. Neurotherapeutics. 2008 Jan;5(1):86-99. doi: 10.1016/j.nurt.2007.10.066. PMID 18164487
- [Result] Finnerup NB, Sindrup SH, Jensen TS. Recent advances in pharmacological treatment of neuropathic pain. F1000 Med Rep. 2010 Jul 14;2:52. doi: 10.3410/M2-52. PMID 21170362
- [Result] Foreman RD, Linderoth B. Neural mechanisms of spinal cord stimulation. Int Rev Neurobiol. 2012;107:87-119. doi: 10.1016/B978-0-12-404706-8.00006-1. PMID 23206679
- [Result] Fruhstorfer H, Gross W, Selbmann O. von Frey hairs: new materials for a new design. Eur J Pain. 2001;5(3):341-2. doi: 10.1053/eujp.2001.0250. PMID 11558991
- [Result] Heinricher MM, Tavares I, Leith JL, Lumb BM. Descending control of nociception: Specificity, recruitment and plasticity. Brain Res Rev. 2009 Apr;60(1):214-25. doi: 10.1016/j.brainresrev.2008.12.009. Epub 2008 Dec 25. PMID 19146877
- [Result] Kalra A, Urban MO, Sluka KA. Blockade of opioid receptors in rostral ventral medulla prevents antihyperalgesia produced by transcutaneous electrical nerve stimulation (TENS). J Pharmacol Exp Ther. 2001 Jul;298(1):257-63. PMID 11408550
- [Result] Kendall NA. Psychosocial approaches to the prevention of chronic pain: the low back paradigm. Baillieres Best Pract Res Clin Rheumatol. 1999 Sep;13(3):545-54. doi: 10.1053/berh.1999.0044. PMID 10562385
- [Result] MENDELL LM, WALL PD. RESPONSES OF SINGLE DORSAL CORD CELLS TO PERIPHERAL CUTANEOUS UNMYELINATED FIBRES. Nature. 1965 Apr 3;206:97-9. doi: 10.1038/206097a0. No abstract available. PMID 14334366
- [Result] Klein T, Magerl W, Hopf HC, Sandkuhler J, Treede RD. Perceptual correlates of nociceptive long-term potentiation and long-term depression in humans. J Neurosci. 2004 Jan 28;24(4):964-71. doi: 10.1523/JNEUROSCI.1222-03.2004. PMID 14749441
- [Result] Kregel J, van Wilgen CP, Zwerver J. Pain assessment in patellar tendinopathy using pain pressure threshold algometry: an observational study. Pain Med. 2013 Nov;14(11):1769-75. doi: 10.1111/pme.12178. Epub 2013 Jun 26. PMID 23802873
- [Result] Ng DT, Spear ED, Walter P. The unfolded protein response regulates multiple aspects of secretory and membrane protein biogenesis and endoplasmic reticulum quality control. J Cell Biol. 2000 Jul 10;150(1):77-88. doi: 10.1083/jcb.150.1.77. PMID 10893258
- [Result] Ochoa JL. Pain mechanisms in neuropathy. Curr Opin Neurol. 1994 Oct;7(5):407-14. doi: 10.1097/00019052-199410000-00008. PMID 7804461
- [Result] Randic M, Jiang MC, Cerne R. Long-term potentiation and long-term depression of primary afferent neurotransmission in the rat spinal cord. J Neurosci. 1993 Dec;13(12):5228-41. doi: 10.1523/JNEUROSCI.13-12-05228.1993. PMID 8254370
- [Result] Sdrulla AD, Xu Q, He SQ, Tiwari V, Yang F, Zhang C, Shu B, Shechter R, Raja SN, Wang Y, Dong X, Guan Y. Electrical stimulation of low-threshold afferent fibers induces a prolonged synaptic depression in lamina II dorsal horn neurons to high-threshold afferent inputs in mice. Pain. 2015 Jun;156(6):1008-1017. doi: 10.1097/01.j.pain.0000460353.15460.a3. PMID 25974163
- [Result] Sjolund B. The ventral spino-olivocerebellar system in the cat. V. Supraspinal control of spinal transmission. Exp Brain Res. 1978 Nov 15;33(3-4):509-22. doi: 10.1007/BF00235571. PMID 215435
- [Result] RaviChandran N, Aw KC, McDaid A. Characterizing the Motor Points of Forearm Muscles for Dexterous Neuroprostheses. IEEE Trans Biomed Eng. 2020 Jan;67(1):50-59. doi: 10.1109/TBME.2019.2907926. Epub 2019 Mar 28. PMID 30932826
- [Result] Rolke R, Magerl W, Campbell KA, Schalber C, Caspari S, Birklein F, Treede RD. Quantitative sensory testing: a comprehensive protocol for clinical trials. Eur J Pain. 2006 Jan;10(1):77-88. doi: 10.1016/j.ejpain.2005.02.003. PMID 16291301
- [Result] Russo CM, Brose WG. Chronic pain. Annu Rev Med. 1998;49:123-33. doi: 10.1146/annurev.med.49.1.123. PMID 9509254
- [Result] Svendsen F, Rygh LJ, Gjerstad J, Fiska A, Hole K, Tjolsen A. Recording of long-term potentiation in single dorsal horn neurons in vivo in the rat. Brain Res Brain Res Protoc. 1999 Jul;4(2):165-72. doi: 10.1016/s1385-299x(99)00018-5. PMID 10446411
- [Result] Sandkuhler J. Learning and memory in pain pathways. Pain. 2000 Nov;88(2):113-118. doi: 10.1016/S0304-3959(00)00424-3. No abstract available. PMID 11050365
- [Result] Sandkuhler J, Liu X. Induction of long-term potentiation at spinal synapses by noxious stimulation or nerve injury. Eur J Neurosci. 1998 Jul;10(7):2476-80. doi: 10.1046/j.1460-9568.1998.00278.x. PMID 9749775
- [Result] Schaible HG. Peripheral and central mechanisms of pain generation. Handb Exp Pharmacol. 2007;(177):3-28. doi: 10.1007/978-3-540-33823-9_1. PMID 17087118
- [Result] Shay BL, Hochman S. Serotonin alters multi-segmental convergence patterns in spinal cord deep dorsal horn and intermediate laminae neurons in an in vitro young rat preparation. Pain. 2002 Jan;95(1-2):7-14. doi: 10.1016/s0304-3959(01)00364-5. PMID 11790462
- [Result] Sivilotti LG, Thompson SW, Woolf CJ. Rate of rise of the cumulative depolarization evoked by repetitive stimulation of small-caliber afferents is a predictor of action potential windup in rat spinal neurons in vitro. J Neurophysiol. 1993 May;69(5):1621-31. doi: 10.1152/jn.1993.69.5.1621. PMID 8389833
- [Result] Smits H, van Kleef M, Holsheimer J, Joosten EA. Experimental spinal cord stimulation and neuropathic pain: mechanism of action, technical aspects, and effectiveness. Pain Pract. 2013 Feb;13(2):154-68. doi: 10.1111/j.1533-2500.2012.00579.x. Epub 2012 Jul 11. PMID 22780956
- [Result] Somers DL, Clemente FR. Contralateral high or a combination of high- and low-frequency transcutaneous electrical nerve stimulation reduces mechanical allodynia and alters dorsal horn neurotransmitter content in neuropathic rats. J Pain. 2009 Feb;10(2):221-9. doi: 10.1016/j.jpain.2008.08.008. Epub 2008 Nov 17. PMID 19010735
- [Result] Stevanato G, Devigili G, Eleopra R, Fontana P, Lettieri C, Baracco C, Guida F, Rinaldo S, Bevilacqua M. Chronic post-traumatic neuropathic pain of brachial plexus and upper limb: a new technique of peripheral nerve stimulation. Neurosurg Rev. 2014 Jul;37(3):473-79; discussion 479-80. doi: 10.1007/s10143-014-0523-0. Epub 2014 Feb 21. PMID 24558032
- [Result] Telles JD, Gabanela Schiavon MA, Rampazo da Silva EP, Liebano RE. Transcutaneous electrical nerve stimulation and cervical joint manipulation on pressure pain threshold. Pain Manag. 2018 Jul 1;8(4):263-269. doi: 10.2217/pmt-2017-0069. Epub 2018 Jun 1. PMID 29856269
- [Result] Treede RD. Gain control mechanisms in the nociceptive system. Pain. 2016 Jun;157(6):1199-1204. doi: 10.1097/j.pain.0000000000000499. PMID 26817644
- [Result] Tompra N, van Dieen JH, Coppieters MW. Central pain processing is altered in people with Achilles tendinopathy. Br J Sports Med. 2016 Aug;50(16):1004-7. doi: 10.1136/bjsports-2015-095476. Epub 2015 Dec 23. PMID 26701922
- [Result] Von Frey M (1896). Untersuchung und ̈ber die Sinnesfunktionen der menschlichen Haut. Erste Abhandlung: Druckempfindung und Schmerz. Abhandlungen der mathematischphysischen Klasse der Königlichen Sa ̈chsischen Gesellschaft der Wissenschaften;. p. 23.
- [Result] Weinstein S (1968). Intensive and extensive aspects of tactile sensitivity as a function of body part, sex, and laterality. In: Kenshalo D, Springfield R, Thomas C, editors. The skin senses. p. 195- 222.
- [Result] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Result] Yang F, Zhang C, Xu Q, Tiwari V, He SQ, Wang Y, Dong X, Vera-Portocarrero LP, Wacnik PW, Raja SN, Guan Y. Electrical stimulation of dorsal root entry zone attenuates wide-dynamic-range neuronal activity in rats. Neuromodulation. 2015 Jan;18(1):33-40; discussion 40. doi: 10.1111/ner.12249. Epub 2014 Oct 10. PMID 25308522
- [Result] Ylinen J. Pressure algometry. Aust J Physiother. 2007;53(3):207. doi: 10.1016/s0004-9514(07)70032-6. No abstract available. PMID 17899675
- [Result] Shacklock M. (2007). Neurodinámica clínica: un nuevo sistema de tratamiento musculoesquelético. Madrid: Elsevier.
- [Result] Amer-Cuenca, J. J. (2010). Programación y aplicación de la estimulación nerviosa eléctrica transcutánea (TENS): guía de práctica clínica basada en la evidencia. Fisioterapia, 32(6), 271-278.